CLINICAL TRIAL: NCT01995448
Title: Prognostic Interest of Leucocyte Immunophenotyping Using Multiparameter 8-color Flow Cytometry During the Acute Phase of Sepsis
Brief Title: Prognostic Interest of Leucocyte Immunophenotyping During the Acute Phase of Sepsis
Acronym: SEPTIFLUX2
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I11020 SEPTIFLUX 2
Record Dates: First submitted 2013-11-15; First posted 2013-11-26 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2015-08

CONDITIONS: Sepsis With Acute Organ Dysfunction
Keywords: The acute phase of Sepsis; multiparameter 8-color flow cytometry
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residue of blood further to NFS.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SEPSIS Blood test: Patient with two criteria of systemic inflammatory response syndrome and a progressive infection which is clinically or microbiologically documented.
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — Residue of blood further to NFS.

SUMMARY:
Septic shock is still a major cause of death in ICU. Sepsis diagnosis is linked with many clinical, hemodynamic and biological criteria which have a low sensitivity and specificity if they are considered separately. The extensive experimental data which have been published contrast with the hematological data collected by the physician at patient's bedside especially regarding neutrophils and platelets levels. When there is no obvious clinical sign, a biological tool reflecting the patient's immune status could be useful to understand the physiopathology of Sepsis and to predict the progression of the disease in the patient. On the long-term it could also help to define management strategies.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years old
* Patient with two criteria of systemic inflammatory response syndrome and a progressive infection which is clinically or microbiologically documented

Exclusion Criteria:

* Pregnancy,
* progressive solid cancer,
* HIV infection,
* history of blood or inflammatory disease,
* long-term immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with two criteria of systemic inflammatory response syndrome and a progressive infection which is clinically or microbiologically documented
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
expression of the marker CD10 | 28 days
  Expression of CD10 on granulocytes.

SECONDARY OUTCOMES:
Progession of SOFA score | 48 hours
Expression of the marker CD16 | 28 days
  Expression of CD16 on granulocytes and on monocytes.
Expression of the marker CD24 | 28 days
  Expression of CD24 on granulocytes.
Expression of the marker CD64 | 28 days
  Expression of CD64 on granulocytes.
Expression of the marker CD14 | 28 days
  Expression of CD14 on monocytes.
Expression of the marker CD3 | 28 days
  Expression of CD3 on T lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FRANCOIS, MD, Principal Investigator — CHU LIMOGES
Locations (9):
- France (9):
  - CHU Bordeaux - Service Réanimation Médicale, Bordeaux
  - CHU Henri MONDOR - Service Réanimation, Créteil
  - CHU Dijon - Service Réanimation Médicale, Dijon
  - CHU Limoges - Service de réanimation polyvalente, Limoges
  - CHU Orléans - Service de Réanimation Médicale, Orléans
  - Hôpital Cochin - service de Réanimation, Paris
  - CHU Poitiers - Service Réanimation, Poitiers
  - CHU Rennes - service de Réanimation, Rennes
  - CHU Tours - Service de Réanimation, Tours

REFERENCES:
- [Derived] Daix T, Guerin E, Tavernier E, Mercier E, Gissot V, Herault O, Mira JP, Dumas F, Chapuis N, Guitton C, Bene MC, Quenot JP, Tissier C, Guy J, Piton G, Roggy A, Muller G, Legac E, de Prost N, Khellaf M, Wagner-Ballon O, Coudroy R, Dindinaud E, Uhel F, Roussel M, Lafon T, Jeannet R, Vargas F, Fleureau C, Roux M, Allou K, Vignon P, Feuillard J, Francois B; Septiflux Trial Group. Multicentric Standardized Flow Cytometry Routine Assessment of Patients With Sepsis to Predict Clinical Worsening. Chest. 2018 Sep;154(3):617-627. doi: 10.1016/j.chest.2018.03.058. Epub 2018 Apr 26. PMID 29705219